CLINICAL TRIAL: NCT01287000
Title: Gulf STUDY: Gulf Long-Term Follow-Up Study
Brief Title: Gulf Long-Term Follow-Up Study
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911076; 11-E-N076
Record Dates: First submitted 2011-01-25; First posted 2011-02-01 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-12-08

CONDITIONS: Cardiovascular Disease; Hematologic Diseases; Immunologic Disease; Cancer; Respiratory Function
Keywords: Respiratory Health Outcomes; Mental Health; Dispersant(s); Oil Spill; Cancer; Natural History
MeSH Terms: conditions — Cardiovascular Diseases; Hematologic Diseases; Immune System Diseases; Neoplasms; Respiratory Aspiration; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Workers and volunteers engaged or potentially engaged in oil spill clean-up operations in the Gulf of Mexico

SUMMARY:
Background:

* There has been little research on the long-term health effects from oil spills, even though at least 10 percent of all oil tanker spills between 1970 and 2009 have affected coastal populations. The Deepwater Horizon disaster, with its release of approximately 5 million barrels (~680,000 tons) of crude oil into the Gulf of Mexico, is far larger than any of the individual tanker spills. Given the magnitude of this spill and the scope of the potential exposures, including the 55,000 workers involved in clean-up efforts and countless residents of the affected areas, researchers are interested in monitoring Gulf clean-up workers to understand the adverse consequences of oil spills in general.
* The Gulf Long-term Follow-up Study will investigate health effects associated with the clean-up activities following the Deepwater Horizon disaster in the Gulf of Mexico on April 20, 2010. More than 100,000 persons completed safety training in preparation for participation in clean-up activities related to the spill. Many of these individuals participated in active clean-up efforts, but others did not. Exposures among persons involved in clean-up range from negligible to potentially significant, especially for workers involved in tasks associated with direct exposure to crude or burning oil, or to chemical dispersants. However, prediction of adverse health effects is not possible because the long-term human health consequences of oil spills are largely unknown. In addition to the oil itself, the widespread economic and lifestyle disruption caused by the oil spill may contribute to mental health problems among this population.

Objectives:

- To investigate potential short- and long-term health effects associated with clean-up activities and exposures surrounding the Deepwater Horizon oil spill.

Eligibility:

- English-, Spanish-, and Vietnamese-speaking workers and volunteers at least 21 years of age engaged or potentially engaged in oil spill clean-up operations in the Gulf of Mexico, or who lived in affected areas (Louisiana, Mississippi, Alabama, and Florida coastal regions).

Design:

* Participants will be divided into groups of those who performed oil-spill clean-up-related work ( exposed ) and those who did not engage in clean-up-related work ( unexposed controls).
* Participants will be screened with a full medical history and physical examination, as well as an interview to determine the nature of their potential exposure.
* Participants will provide blood, hair, toenail, urine, and saliva (spit) samples. Participants may also have a lung function exam.
* Participants will have researchers collect dust from their homes by using wipes and special vacuum bags.
* Participants will also provide detailed contact information, including their Social Security number, to be contacted in the future for long-term health follow-up appointments. These appointments will include 30-minute telephone interviews every 2 years.

DETAILED DESCRIPTION:
The Gulf Long-term Follow-up Study (GuLF STUDY) will investigate potential short- and long-term health effects associated with the clean-up activities following the Deepwater Horizon disaster in the Gulf of Mexico on April 20, 2010. Crude oil, burning oil, and the dispersants used during clean-up efforts contain a range of known and suspected toxins. Over 100,000 persons have completed safety training in preparation for participation in clean-up activities related to the spill. While many of these individuals participated in active clean-up efforts, others did not. Exposures among persons involved in clean-up range from negligible to potentially significant, especially for workers involved in tasks associated with direct exposure to crude or burning oil, or to chemical dispersants. However, prediction of adverse health effects is not possible because the long-term human health consequences of oil spills are largely unknown due to the dearth of research in this area. The potential health effects associated with the levels of exposure experienced by clean-up workers are largely unstudied. Heat and stress experienced by these workers may also have adverse long-term health effects. In addition to the oil itself, the widespread economic and lifestyle disruption caused by the oil spill may contribute to mental health problems among this population.

The over-arching hypotheses of this study are:

1. Exposure to constituents of oil, dispersants, and oil-dispersant mixtures, and to spill-related stress by workers engaged in clean-up of the Deepwater Horizon oil spill are associated with adverse health effects, particularly respiratory, neurological, hematologic, and psychological or mental health.
2. There are exposure-response relationships between the above exposures and health effects.
3. Biomarkers of potentially adverse biologic effects are associated with the above exposures.

Based on what is known about individuals involved in clean-up efforts, the cohort will consist primarily of English-, Spanish-, or Vietnamese-speaking adults who performed oil-spill clean-up-related work ( exposed ) and similar persons who did not engage in clean-up-related work ( unexposed controls). Accommodations for enrolling participants speaking other languages will be developed through community collaborations as appropriate. Workers will be sampled from across job/potential exposure groups. A total of approximately 55,000 persons are expected to be enrolled into the cohort. A random sample of the full cohort, stratified by category of job/potential exposure (including N~6,000 with no oil-spill work to serve as controls) and oversampled for workers with higher potential exposures, will be enrolled into an Active Follow-up Sub-cohort (N~20,000). A random sample of the Active Follow-up Sub-cohort, also stratified by category of job/potential exposure and oversampled for workers with higher potential exposures, will be enrolled into a Biomedical Surveillance Sub-cohort (N~5,000). Participants will be interviewed about their clean-up-related tasks, demographic and socioeconomic factors, occupational and health histories, psychosocial factors, and physical and mental health. Members of the Active Follow-up Sub-cohort will also be asked to provide biological samples (blood, urine, hair, toenail clippings, and possibly saliva) and environmental samples (house dust) and will have basic clinical measurements (height, weight, waist and hip circumference, blood pressure, urinary glucose levels, FEV1 and FVC as a measure of pulmonary function) taken during home visits at baseline. The Biomedical Surveillance Sub-cohort will participate in a more comprehensive clinical assessment after the initial home visit, including more comprehensive pulmonary function testing, neurological testing, and collection of additional biological and environmental samples. The specific tests to be performed and clinical protocols will be developed in collaboration with extramural investigators selected through a request for proposals (RFP). When developed, the protocol for this portion of the study will be submitted separately to the Institutional Review Board as a study amendment.

Exposures will be estimated using detailed job-exposure matrices developed from data from monitoring performed by different agencies and organizations during the crisis, as well as information on recommended or actual use of personal protection, information obtained by interview, and the available scientific literature. It should be noted that, in the absence of individual or group monitoring data for most workers, estimates of exposure, whether based on job activities or on more refined job-exposure matrices, will indicate the degree of potential exposure (i.e., exposure opportunity) rather than known exposure. We will investigate acute health effects via self-report from the enrollment interview among all cohort members and also via clinical measures and biological samples from Active Follow-up Sub-cohort members. All cohort members will be followed for development of a range of health outcomes through record linkage (cancer, mortality) and if feasible, through linkage with electronic medical records that may become available during the course of follow-up. Health outcomes among the Active Follow-up Sub-cohort will also be identified through self-report via periodic follow-up interviews. Additional outcome information will be obtained on the Biomedical Surveillance Sub-cohort from periodic follow-up clinical evaluations (e.g., spirometry, neurological testing) and analysis of follow-up biospecimens (e.g., immunologic parameters, liver function, renal function, DNA damage). Follow-up of the entire cohort is initially planned for 10 years, with extended follow-up possible depending upon scientific and public health needs and the availability of funds.

Recruitment of subjects should begin in March 2011, with the telephone interviews expected to be completed within 12-24 months and the baseline home visits within 18-26 months. For the home visits, we will initially target workers residing in the four most affected Gulf States (LA, MS, AL, and FL), although we may expand to other states if further information about the geographic distribution of workers and their potential exposures warrants additional follow-up in these states. We will work closely with a Community Advisory Board to develop community support for this study and appropriate communications and study materials.

ELIGIBILITY:
* INCLUSION CRITERIA:

We anticipate screening as many as 90,000 individuals in order to recruit approximately 55,000 volunteers primarily from the four most affected Gulf States* (LA, MS, AL, and FL) into the cohort, which will include a randomly sampled Active Follow-up Sub-cohort of approximately 24,000 individuals nested within it. Eligibility criteria for the cohort include:

* 21 years of age or older
* Fall into one of two oil-related exposure categories:

  * Potentially exposed subjects must have completed at least one day of oil-spill clean-up-related work (other than safety training), either paid or volunteer.
  * Unexposed subjects will be individuals who were not directly involved in oil spill clean-up activities, but who worked near the oil spill or completed some oil spill worker training.
* Unexposed subjects will be individuals who were not directly involved in oil spill clean-up activities, but who worked near the oil spill or completed some oil spill worker training.
* pregnant women will be allowed to enroll in the study, and women who become pregnant during the study will not be withdrawn.

EXCLUSION CRITERIA:

* Children will not be enrolled because they were not allowed to participate in clean-up activities.
* Those who were deemed medically ineligible to participate in clean-up activities because of pre-existing conditions are excluded because they won t be representative of those individuals who were engaged in clean-up activities.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Workers and volunteers engaged or potentially engaged in oil spill clean-up operations in the Gulf of Mexico
Sampling Method: Non-Probability Sample
Enrollment: 32658 (Actual)
Dates: Start 2011-03-24 (Actual)

PRIMARY OUTCOMES:
To investigate potential short- and long-term health effects associated with oil spill clean-up activities/exposures surrounding the Deepwater Horizon Disaster. | Ongoing
  To investigate potential short- and long-term health effects associated with oil spill clean-up activities/exposures surrounding the Deepwater Horizon Disaster.

SECONDARY OUTCOMES:
To investigate biomarkers of potentially adverse biological effect in relation to oil spill clean-up activities/exposures. | Ongoing
  To investigate biomarkers of potentially adverse biological effect in relation to oil spill clean-up activities/exposures.

CONTACTS AND LOCATIONS:
Overall Officials: Dale P Sandler, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- Social & Scientific Systems, Durham, North Carolina, United States